# Impacts of Alcohol Warning Labels: an Online Experiment

NCT number NCT06442800 Document Date 06/28/2024 Consent Form Version Date: June 28, 2024

**IRB Study** # 23-1218

**Title of Study**: Developing New Labels **Principal Investigator**: Marissa Hall

Principal Investigator Department: Health Behavior Principal Investigator Phone Number: (919) 445-1310 Principal Investigator Email Address: mghall@unc.edu

Funding Source and/or Sponsor: NIH National Institute on Alcohol Abuse and Alcoholism

Concise Summary. We would like to invite you to take part in a brief research study to better understand people's thoughts and perceptions about alcohol labels. This survey is open to U.S. residents aged 21 or older who consume alcohol. The study will involve a one-time computer survey about your reactions to alcohol messages, lasting about 15 minutes. We will also collect some personal information that will be separated from your survey responses and will never be published or shared. The two potential risks to participating in this study include (1) discomfort while answering the survey and (2) loss of privacy resulting from accidental disclosure of responses to survey questions. Not only are these risks small, but the risk of a rare accidental disclosure would also be small. We do not anticipate any direct benefits from participation.

#### What are some general things you should know about research studies?

You are being asked to take part in a research study. To join the study is voluntary. You may choose not to participate, or you may withdraw your consent to be in the study, for any reason, without penalty.

### What is the purpose of this study?

The purpose of this research study is to study reactions to labels on alcohol products. About 1,000 participants will take part in the study.

# How long will your part in this study last?

You will be in the study for about 10-15 minutes. This will be a one-time survey about your thoughts and perceptions about labels on alcohol products with no follow-up expected.

## What are the possible benefits from being in this study?

Research is designed to benefit society by gaining new knowledge. There is little chance you will benefit from being in this research study.

#### What are the possible risks or discomforts involved from being in this study?

The two potential risks to participating in this study include (1) feeling uncomfortable while answering the survey questions and (2) loss of privacy resulting from accidental disclosure of responses to survey questions. Not only are these risks small, but the risk of a rare accidental disclosure would also be small because we are not collecting sensitive information.

#### How will information about you be protected?

Some personal identifying information (such as name, sex assigned at birth, birthdate, and city of birth) will be collected during this survey. This information will <u>never</u> be published or shared alongside any research findings. It will only be used to create a randomly generated code for your data which will no longer be tied to any personal information. Your responses to the survey questions will be kept confidential. Participants will not be identified in any report or publication about this study. We may use de-identified data from this study in future research without additional consent. A de-identified version of the dataset may be made available publicly online.

Although every effort will be made to keep research records private, there may be times when federal or state law requires the disclosure of such records, including personal information. This is very unlikely, but if disclosure is ever required, UNC-Chapel Hill will take steps allowable by law to protect the privacy of personal information.

## Will you save my research data to use in future research studies?

Deidentified data from this study will be submitted to the National Institute of Mental Health Data Archive. Deidentified information means that all personal information about research participants such as name, address, and phone number is removed and replaced with a code number. This data archive allows researchers to collect and share deidentified information with each other. It is a large database where information from many studies is stored and managed.

## What is a Certificate of Confidentiality?

This research is covered by a Certificate of Confidentiality. With this Certificate, the researchers may not disclose or use information, or documents that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings in the United States, for example, if there is a court subpoena, unless you have consented for this use.

The Certificate cannot be used to refuse a request for information from personnel of a federal or state agency that is sponsoring the study for auditing or evaluation purposes. The Certificate of Confidentiality will not be used if disclosure is for other scientific research, as allowed by federal regulations protecting research subjects or for any purpose you have consented to in this informed consent document.

You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

#### What if you want to stop before your part in the study is complete?

You can withdraw from this study at any time, without penalty. You can skip survey questions for any reason, and you will receive payment even if you skip questions.

#### Will you receive anything for being in this study?

Upon completion of the 10-15 minute survey, you will receive compensation in the reward type and amount that you have agreed to with the platform through which you entered this survey.

## What if you have questions about this study?

You have the right to ask, and have answered, any questions you may have about this research. Contact the Principal Investigator listed above with any questions, complaints, or concerns you may have.

## What if you have questions about your rights as a research participant?

All research on human volunteers is reviewed by a committee that works to protect your rights and welfare. If you have questions or concerns about your rights as a research subject, or if you would like to obtain information or offer input, you may contact the Institutional Review Board at 919-966-3113 or by email to <a href="mailto:IRB\_subjects@unc.edu">IRB\_subjects@unc.edu</a>.

By continuing to the survey below, you acknowledge that you have read and understand the information on this page and agree to be in this research study. Thank you!